CLINICAL TRIAL: NCT03828955
Title: Evaluation of Soybean Peptides Product on Regulation of Blood Pressure Effect by Clinical Trial
Brief Title: Evaluation of Soybean Peptides Product on Regulation of Blood Pressure Effect in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, School of Health Diet and Industry Managment, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CS15123
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: soybean peptides; clinical trial; blood preesure; SBP; DBP
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soybean peptides (Experimental): Subjects receive two bags soybean peptides per day for 8 weeks of a stage.
  Interventions: Dietary Supplement: Soybean peptides
- Placebo (Placebo Comparator): Subjects receive two bags starch placebo of similar appearance per day for 8 weeks of a stage.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soybean peptides — Subjects receive two bags soybean peptides per day for 8 weeks of a stage. Anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), body weight, body fat, waistline, hipline and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST and ALT were measured every four weeks.
  Arms: Soybean peptides
Dietary Supplement: Placebo — Subjects receive two bags of starch placebo of similar appearance per day for 8 weeks of a stage. Anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), body weight, body fat, waistline, hipline, and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST, and ALT were measured every four weeks.
  Arms: Placebo

SUMMARY:
This is the report to assess supplementation with soybean peptides on blood pressure among people with mild hypertension. Overall, soybean peptide consumption for 8 weeks could successfully reduce mean diastolic and systolic BP through the suppression of Angiotensin-converting enzyme (ACE) linked to downstream suppression of angiotensin II formation, which further decreases the sympathetic outflow that leads to hypertension.

DETAILED DESCRIPTION:
This is the report to assess supplementation with soybean peptides on blood pressure among people with mild hypertension. Thirty subjects with systolic blood pressure (SBP) between 120 and 159 mm Hg and/or diastolic blood pressure (DBP) between 80 and 99 mm Hg were randomized to ingest 2 bags of soybean peptides or placebo per day for 8 weeks of a stage. Anthropometric measurements (blood pressure, body weight, body fat) and blood biochemical markers including fasting blood glucose (FBG), albumin, total cholesterol (TC), triglyceride (TG), HDL-C, LDL-C, creatinine (Cr), blood urea nitrogen (BUN), AST, ALT) were examined every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were untreated hypertensive men or women aged between 20 and 80 years old with SBP between 120 and 159 mmHg and/or DBP between 80 and 99 mmHg as measured in a sitting position

Exclusion Criteria:

* Subjects were excluded if they had a history of major cardiovascular disease or severe liver dysfunction;
* Diastolic blood pressure ≥ 100 mmHg or Systolic blood pressure ≥ 160 mmHg;
* Alcoholic;
* US-controlled diabetics;
* Stoke in past one year;
* Mental diseases or melancholia;
* Pregnancy or breast-feeding a child;
* Renal dysfunction;
* Allergic to Soybean peptides.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The soy bean peptides anti-hypertensive measure blood pressure (SBP and DBP) | 8 weeks
  values chang of systolbbic and diastolic BPs between before to after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

REFERENCES:
- [Background] Lo WM, Li-Chan EC. Angiotensin I converting enzyme inhibitory peptides from in vitro pepsin-pancreatin digestion of soy protein. J Agric Food Chem. 2005 May 4;53(9):3369-76. doi: 10.1021/jf048174d. PMID 15853374
- [Background] Rizzello CG, Cassone A, Di Cagno R, Gobbetti M. Synthesis of angiotensin I-converting enzyme (ACE)-inhibitory peptides and gamma-aminobutyric acid (GABA) during sourdough fermentation by selected lactic acid bacteria. J Agric Food Chem. 2008 Aug 27;56(16):6936-43. doi: 10.1021/jf800512u. Epub 2008 Jul 16. PMID 18627167
- [Background] Yoshiji H, Kuriyama S, Fukui H. Angiotensin-I-converting enzyme inhibitors may be an alternative anti-angiogenic strategy in the treatment of liver fibrosis and hepatocellular carcinoma. Possible role of vascular endothelial growth factor. Tumour Biol. 2002 Nov-Dec;23(6):348-56. doi: 10.1159/000069792. PMID 12677092